CLINICAL TRIAL: NCT03338569
Title: Evaluating Vitamin C in Septic Shock: A Randomized Double Blind Placebo Controlled Trial
Brief Title: Vitamin C and Septic Shock
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00000625
Record Dates: First submitted 2017-10-31; First posted 2017-11-09 (Actual); Results first posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Septic Shock; Sepsis
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Sham Comparator): Placebo designed to mimic intervention
  Interventions: Drug: Placebo
- Intervention (Active Comparator): 6000 mg per day Vitamin C supplement
  Interventions: Drug: Vitamin C

INTERVENTIONS:
Drug: Vitamin C — Continuous infusion of vitamin C
  Other Names: ascorbic acid
  Arms: Intervention
Drug: Placebo — Placebo designed to mimic intervention
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled clinical trial to compare Vitamin C versus placebo for patients presenting to the ICU with a diagnosis of septic shock.

DETAILED DESCRIPTION:
This is a multi-site, randomized, double-blind, placebo-controlled trial comparing a regimen of moderate-dose (6000 mg per day) Vitamin C supplementation versus placebo for the treatment of patients presenting to the ICU with septic shock. Both groups will continue to receive all other standard of care measures for septic shock as clinically indicated. Groups will be enrolled and receive study drug/placebo for 4 days (96 hours) or until 24 hours post-last pressor dose, whichever is sooner.

ELIGIBILITY:
Inclusion Criteria:

* • Capability to provide written consent from participant or legally authorized representative (LAR) if the participant is unable or incapacitated due to severity of illness.

  * Age ≥ 18 years
  * Septic shock as pragmatically defined as:

    o Order for intravenous antimicrobials with either procalcitonin > 2 mg/dL within 24 hours of enrollment OR other clinical suspicion of infection or confirmed infection AND
  * Hypotension requiring vasopressor therapy, despite fluid resuscitation of at least 30 cc/kg AND
  * Lactate > 2 mmol/L 24 hr prior to enrollment AND
  * Presence of sepsis defined as equal to or greater than 2 SIRS criteria and/or acute increase in qSOFA score of 2 points or more.

    * SIRS criteria: 1) Temperature greater than 38° or less than 36° Celsius. 2) Heart rate greater than 90 beats per minute. 3) Respiratory rate greater than 20 breaths per minute OR arterial carbon dioxide tension less than 32 mmHg. 4) White blood cell count greater than 12,000 cell/µL, less than 4,000 cells/µL, OR band cells greater than 10% of the total white blood cell population.
    * qSOFA: 1 point each is assigned for: 1) systolic blood pressure below 100, 2) respiratory rate greater than 22, and 3) mental status not at baseline.

Exclusion Criteria:

* • Unable to start infusion within 24 hours of septic shock identification

  * Currently pregnant or breastfeeding
  * Patient to receive comfort measures only
  * Cardiac Arrest
  * Cardiovascular Surgery patients receiving prophylactic peri-operative antibiotics < 48 hours post-operation
  * Participation in another study involving an investigational product within 30 days of the baseline visit
  * Allergy to Vitamin C
  * History of nephrolithiasis
  * History of G6PD deficiency
  * ESRD patients, transplant eligible on dialysis currently taking vitamin C supplementation
  * Clinical course that treating clinician decides would preclude safe participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-08-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wacker DA, Burton SL, Berger JP, Hegg AJ, Heisdorffer J, Wang Q, Medcraft EJ, Reilkoff RA. Evaluating Vitamin C in Septic Shock: A Randomized Controlled Trial of Vitamin C Monotherapy. Crit Care Med. 2022 May 1;50(5):e458-e467. doi: 10.1097/CCM.0000000000005427. Epub 2022 Jan 5. PMID 34982738

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Vitamin C
  Vitamin C: Continuous infusion of vitamin C
Period: Overall Study
Arm/Group | Placebo | Intervention
Started | 64 | 61
Completed | 56 | 56
Not Completed | 8 | 5
Not completed — Physician Decision | 8 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Intervention | Total
Number analyzed (Participants) | 64 | 61 | 125
Age, Continuous [Mean (Full Range); unit: years] | 73 [60.7 to 80] | 68.9 [60.1 to 79.9] | 71 [60.1 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 31 | 62
  Male | 33 | 30 | 63
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 59 | 59 | 118
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 64 | 61 | 125

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With ICU Mortality
Description: Outcome is reported as the number of patients who expired while receiving care in the intensive care unit (ICU).
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 64 | 61
Participants | 20 | 14

2. Primary Outcome: All Cause Mortality at 28 Days
Description: Outcome is reported as the number of participants who have expired at 28 days post intervention
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 64 | 61
Participants | 26 | 16

3. Secondary Outcome: Duration of Vasopressor Therapy
Description: Outcome is reported as the duration in hours of vasopressor therapy post intervention administration
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 64 | 61
hours | 27.1 [16.4 to 45.2] | 27.7 [13.6 to 47.6]

4. Secondary Outcome: Duration of ICU Stay Post Intervention Administration
Description: Outcome is reported as the duration (in days) that participants require care in the intensive care unit (ICU) post intervention administration
Time Frame: 28 days
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 64 | 61
days | 2.6 [1.5 to 5.3] | 2.9 [1.8 to 7.5]

5. Secondary Outcome: Time to Lactate Clearance Post Intervention Administration
Time Frame: 28 days
Population: Measure was not collected
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Rate of Lactate Clearance Post Intervention Administration
Description: Outcome is reported as the number of participants who clear lactate from the bloodstream at 24, 48, 72, and 96 hours post intervention. Clearance is defined as a serum concentration of 2.0 mmol/l or less.
Time Frame: 24, 48, 72, and 96 hours post intervention
Population: All participants who completed 96 hours of testing are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 45 | 43
Participants
  24 hours | 13 | 12
  48 hours | 18 | 16
  72 hours | 18 | 18
  96 hours | 19 | 18

7. Secondary Outcome: Rate of Procalcitonin Clearance Post Intervention Administration
Time Frame: 4 days
Population: Outcome was not collected.
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants With Need for Renal Replacement Therapy
Description: Outcome is reported as the number of participants who require renal replacement therapy
Time Frame: 4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 64 | 61
Participants | 2 | 10

9. Secondary Outcome: Change in Serum Creatinine
Description: Outcome is report as the change in serum creatinine between baseline and 4 days following treatment. Outcome is reported in units of mg/dl.
Time Frame: Baseline and 4 days
Population: All participants for whom baseline and 96-hour creatinine data is available are included in this analysis.
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 56 | 49
mg/dl | 0.5 [-0.1 to 0.7] | .4 [0 to 0.7]

10. Secondary Outcome: Change in Sequential Organ Failure Assessment (SOFA) Score
Description: SOFA score is a mortality prediction score that is based on the degree of dysfunction of 6 organ systems. Total scores range from 0 to 24, with higher scores indicating higher likely mortality.
Time Frame: Baseline and 4 days
Population: All participants for whom baseline and 96-hour SOFA scores were available are included in this analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 61 | 58
score on a scale | 4 [2 to 6] | 4 [2 to 6]

11. Secondary Outcome: Change in Acute Physiology and Chronic Health Evaluation (APACHE) Scores
Description: APACHE score is a severity-of-disease classification system that is calculated from a patient's age and 12 routine physiological measurements. Total scores are computed based on several measurements and range from 0 to 71 with higher scores corresponding to more severe disease and a higher risk of death.
Time Frame: Baseline and 4 days
Population: All participants for whom APACHE scores at baseline and 4 days post intervention were available are included.
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 61 | 58
score on a scale | 7 [1 to 12] | 5 [3 to 10]

12. Secondary Outcome: Total Intravenous Fluid Administered
Description: Outcome is reported as the total volume of intravenous fluid (in liters) administered to participants during 24 hours following the initiation of study treatment.
Time Frame: 24 hours
Population: All participants for whom total intravenous fluid administration data was available are included.
Measure: Mean (Inter-Quartile Range); unit: liters
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 64 | 60
liters
  6 hours post initiation of study treatment | .76 [.36 to 1.26] | 1.07 [.72 to 1.64]
  24 hours post initiation of study treatment | 3.37 [1.98 to 4.7] | 3.59 [2.52 to 5.02]

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Placebo | Intervention
All-Cause Mortality (participants affected / at risk) | 26/64 | 16/61
Serious Adverse Events (participants affected / at risk) | 3/64 | 4/61
Other Adverse Events (participants affected / at risk) | 9/64 | 8/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=64) | Intervention (N=61)
Elevated Troponin w/o ST elevation (Cardiac disorders) | 0 (0) | 2 (2)
New or worsening heart failure (Cardiac disorders) | 2 (2) | 0 (0)
Arrythmia (Cardiac disorders) | 1 (1) | 0 (0)
Bleeding (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=64) | Intervention (N=61)
Loose stools (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
New or worsening heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Arrythmia (Cardiac disorders) | 3 (3) | 4 (7)
Elevated Troponin w/o ST elevation (Cardiac disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Bleeding event (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Maculopapular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/69/NCT03338569/Prot_SAP_001.pdf
  • Informed Consent Form (2020-01-23): https://cdn.clinicaltrials.gov/large-docs/69/NCT03338569/ICF_002.pdf